CLINICAL TRIAL: NCT04301336
Title: Comparative Effectiveness of the Different Treatment Modalities for Management of Vaso-occlusive Painful Crisis in Pediatric Sickle Cell Disease
Brief Title: Different Treatment Modalities in the Management of the Painful Crisis in Pediatric Sickle- Cell Anemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Benisuef university hospital (Unknown); University of Arizona (Other); Maternity and Children Hospital, Makkah (Other)
Responsible Party: Principal Investigator, SHAIMAA MAHMOUD NASHAT SHAYED ABDELHALIM, Dr.Shaimaa Mahmoud Nashat Sayed Abdelhalim, Ph.D. Researcher and Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Novel TTT of pedia VOC/SCA
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Vaso-occlusive Crisis; Sickle Cell Disease; Sickle Cell Anemia in Children
Keywords: omega3; Vaso-occlusive painful crisis; Pediatric sickle cell anemia; comparative effective analysis in VOC; Anti-inflammatory effect of Vit-D; Anti-hemolytic effect of Vit-D; Anti-hyperlipidemia of Vit-D; effect of omega-3 on blood rheology; effect of omega-3 on blood viscosity; Antiaggregation effect of omega-3; Anti-inflammatory effect of statins; Anti-inflammatory effect of zinc supplements; effect of zinc supplements on blood viscosity; effect of zinc supplements on blood rheology; Antiaggregation effect of zinc supplements; pediatric sickle cell disease
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell | interventions — Docosahexaenoic Acids; Zinc Sulfate; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Cardiovascular Agents; Simvastatin; Hydroxyurea; Morphine

STUDY DESIGN:
Intervention Model Description: Four experimental groups, one control group
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Omega-3 experimental group (Experimental): 50 patients from each participating hospital that will receive Omega-3 supplementation (300-400mg EPA & 200-300mg DHA) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Interventions: Drug: Omega 3; Drug: Hydroxy Urea; Drug: Folic Acid Supplementation; Drug: Morphine Sulfate; Procedure: blood transfusion session
- Vit-D experimental group (Experimental): 50 patients from each participating hospital that will receive Vit-D medication (1500 IU to 3500 IU ) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Interventions: Drug: Vit D; Drug: Hydroxy Urea; Drug: Folic Acid Supplementation; Drug: Morphine Sulfate; Procedure: blood transfusion session
- Zinc supplements experimental group (Experimental): 50 patients from each participating hospital that will receive Zinc supplements (15 mg to 50 mg ) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Interventions: Drug: Zinc sulfate; Drug: Hydroxy Urea; Drug: Folic Acid Supplementation; Drug: Morphine Sulfate; Procedure: blood transfusion session
- Statin experimental group (Experimental): 50 patients from each participating hospital that will receive Simvastatin orally (20 mg to 40 mg ) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Interventions: Drug: Statins (Cardiovascular Agents); Drug: Hydroxy Urea; Drug: Folic Acid Supplementation; Drug: Morphine Sulfate; Procedure: blood transfusion session
- Ordinary hospital treatment group (Active Comparator): 50 patients from each participating hospital that will receive the ordinary treatment of Hydroxyurea (20 mg/kg/day) with monitoring blood count every 2 weeks maximum daily dose: (40 mg/kg/day) for 8 consecutive months up to 10 months.
  in addition, Folic Acid dose of 0.5 to 1 mg daily for 3 to 4 weeks until definite hematologic response in addition, Morphine medication as a pain killer is administered, if Patient weight <50 kg: Opioid naïve: Initial: 0.05 mg/kg/dose; usual maximum initial dose: 1 to 2 mg/dose.
  This group received regular blood transfusion session.
  Interventions: Drug: Hydroxy Urea; Drug: Folic Acid Supplementation; Drug: Morphine Sulfate; Procedure: blood transfusion session

INTERVENTIONS:
Drug: Omega 3 — Omega-3 supplementation (300-400mg EPA & 200-300mg DHA) per day for 8 consecutive months up to 10 months
  Other Names: omega-3 supplementation capsules
  Arms: Omega-3 experimental group
Drug: Vit D — 50 patients from each participating hospital that will receive Vit-D medication (1500 IU to 3500 IU ) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Other Names: Vit-D medication oral drops
  Arms: Vit-D experimental group
Drug: Zinc sulfate — 50 patients from each participating hospital that will receive Zinc supplements (15 mg to 50 mg ) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Other Names: Zinc tablet medication
  Arms: Zinc supplements experimental group
Drug: Statins (Cardiovascular Agents) — 50 patients from each participating hospital that will receive Simvastatin orally (20 mg to 40 mg ) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of hydroxyurea, Folic acid, pain killer plus regular blood transfusion with a dose de-escalation methods till efficacy of experimental treatment proved.
  Other Names: Simvastatin 20mg
  Arms: Statin experimental group
Drug: Hydroxy Urea — 50 patients from each participating hospital that will receive the ordinary treatment of Hydroxyurea (20 mg/kg/day) with monitoring blood count every 2 weeks maximum daily dose: (40 mg/kg/day) for 8 consecutive months up to 10 months.
  Other Names: Hydroxy Urea tablet medication 20mg/kg/day
Drug: Folic Acid Supplementation — Folic Acid dose of 0.5 to 1 mg daily for 3 to 4 weeks until definite hematologic response
  Other Names: Folic Acid tablet medication 1mg/day
Drug: Morphine Sulfate — Morphine medication as a pain killer is administered, if Patient weight <50 kg: Opioid naïve: Initial: 0.05 mg/kg/dose; usual maximum initial dose: 1 to 2 mg/dose.
  Other Names: Morphine Sulfate intra venous medication
Procedure: blood transfusion session — Regular blood transfusion session based on patient hematological profile starts from one session every 2 weeks.

SUMMARY:
The aim of the present study is comparing the effectiveness of different treatment regimens for investigating the therapeutic potential for each one in management of Vaso-occlusive pain in pediatric sickle cell disease. In addition, investigators apply the Cost-effectiveness analysis (CEA) as a form of economic analysis that compares the relative costs and outcomes (effects) for different treatment regimens on vaso-occlusive painful crisis.

DETAILED DESCRIPTION:
"Sickle cell disease is an inherited blood disorder characterized by defective hemoglobin (a protein in red blood cells that carries oxygen to the tissues of the body).

Sickle cell disease involves the red blood cells, or hemoglobin, and their ability to carry oxygen. Normal hemoglobin cells are smooth, round, and flexible, like the letter "O," so they can move through the vessels in our bodies easily. Sickle cell hemoglobin cells are stiff and sticky and form into the shape of a sickle, or the letter "C," when they lose their oxygen. These sickle cells tend to cluster together and cannot easily move through the blood vessels. The cluster causes a blockage in small arteries or capillaries and stops the movement of healthy, normal oxygen-carrying blood. This blockage is what causes the painful and damaging complications of sickle cell disease".

"Acute vaso-occlusive crisis (VOC) is a hallmark of sickle cell disease (SCD). Multiple complex pathophysiological processes can result in pain during a VOC. Despite significant improvements in the understanding and management of SCD, little progress has been made in the management of pain in SCD, although new treatments are being explored".

The Painful Episodes:

"The day-to-day management of sickle cell disease often equates with the management of acute and chronic pain. Patients manage many painful events at home so that hospital visits underestimate the frequency of pain

Acute painful episodes are the most commonly encountered vaso-occlusive events in patients of all ages. Presumed to be caused by sickle vaso-occlusion, pain often starts in young children as the hand-foot syndrome or dactylitis, a painful swelling of hands and feet due to inflammation of the metacarpal and metatarsal periosteum. Painful episodes, which last from hours to many days, usually occur with little warning and a clear precipitating event is not often found.

ELIGIBILITY:
Inclusion Criteria:

Any case with the full manifestation of sickle cell disease accompanied by acute painful crisis aged from 5-15 years old.

Exclusion Criteria:

1. The presence of any other chronic illness.
2. Patient age>18 years old or < 3 years old.
3. Patients with hepatic diseases including cholestasis hepatic encephalopathy and jaundice.
4. Patients with renal impairment
5. Diabetic patients

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
C-reactive protein mg/L | 10 months
  C-reactive protein milligrams per deciliter
Hematocrit % | 10 months
  Hematocrit level in percentage value
Fibrinogen mg/dl | 10 months
  Fibrinogen concentration in milligrams per deciliter
Total cholesterol Mg/dl | 10 months
  Total cholesterol milligrams per deciliter
HDL cholesterol Mg/dl | 10 months
  HDL cholesterol milligrams per deciliter
LDL cholesterol Mg/dl | 10 months
  LDL cholesterol milligrams per deciliter
Triglycerides Mg/dl | 10 months
  Triglycerides milligrams per deciliter
leukocytes count μl | 10 months
  leukocytes in microliter
hemoglobin (Hbg) g/dL | 10 months
  hemoglobin (Hbg) gram/deciliter
White blood cells count | 10 months
  White blood cells count in a cubic milliliter of blood
Lactic acid dehydrogenase U/L | 10 months
  Lactic acid dehydrogenase unit per litter
Reticulocyte count % | 10 months
  Reticulocyte count percentage
Red blood cell (erythrocyte ) sedimentation rate mm/hr | 10 months
  erythrocyte sedimentation rate in millimeters (mm) per one hour(hr)
lymphocyte count µL | 10 months
  lymphocyte count in 1 microliter (µL) of blood
Granulocyte absolute count cells/microliter | 10 months
  Granulocyte cells numbers in microliter
Granulocytes,percentage (GR, pct) | 10 months
  percentage of white blood cells with granules in percentage

CONTACTS AND LOCATIONS:
Overall Officials: John E. Murphy [Professor of Pharmacy Practice and Science], PharmD, Study Director — University of Arizona, College of Pharmacy; Mohamed H Meabad [Prof of Pediatrics], M.D, Study Director — Beni-Suef University, Faculty of medicine; AHMED A ALBERRY [Assistant prof of clinical pharmacology], M.D, Study Director — Beni-Suef University, Faculty of medicine; RAGHDA R SAYED [Lecturer of Clinical Pharmacy, Ph.D., Study Director — Beni-Suef University, Faculty of Pharmacy; Shaimaa M Nashat Sayed Abdelhalim, Ph.D Student, Principal Investigator — Beni-Suef University, Faculty of Pharmacy; Ahmed F Mahmoud Hussein, MS.c, Study Director — Beni-Suef Health insurance hospital
Locations (4):
- Egypt (3):
  - Faculty of medicine, Beni-suef univeristy - Beni-Seuf university hospital, Banī Suwayf
  - Faculty of Pharmacy, Beni-Suef university, Banī Suwayf
  - Health insurance hospital, Banī Suwayf
- Maternity and Children hospital, Mecca, Saudi Arabia